CLINICAL TRIAL: NCT03540121
Title: Improving Adherence in Kidney Recipients: a Randomized Controlled Trial of a Post-transplant Education Intervention
Brief Title: Video Education and Behaviour Contract to Optimize Adherence in Renal Transplants
Acronym: VECTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Authority - Regina Area (Other); Southern Alberta Transplant Program (Unknown); University of Illinois Health Sciences System (Unknown); American Society of Transplantation Research Network (Unknown); University of Alberta Transplant Recipient Program (Unknown); Vancouver Coastal Health (Other Government); Providence Health, St. Pauls Hospital - Renal Transplant Program (Unknown)
Responsible Party: Principal Investigator, Holly Mansell, Associate Professor, College of Pharmacy and Nutrition, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 99399
Record Dates: First submitted 2018-04-27; First posted 2018-05-30 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Kidney Transplantation; Medication Adherence
Keywords: video; contract; patient education
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video education + adherence contract (Experimental): electronically delivered video education (at transplant discharge) + electronic adherence contract (1 month after enrolment)
  Interventions: Behavioral: Video education + adherence contract
- Standard education (No Intervention): standard of care education provided at each transplant center (control emails will be provided at intervention time points)

INTERVENTIONS:
Behavioral: Video education + adherence contract — Participants will receive standard education along with the home-based video education plus an adherence contract. Following the baseline assessment, access to videos will be provided electronically so that the patient can watch them at home. The videos will be initially viewed in the following order: Video 1: Introduction, Video 2: Medications, Video 3: Your New Life. Approximately one month after transplant, after the video series has been viewed in its entirety, participants will receive an email link inviting participants to reflect on their goals about transplantation and pledging to taking their medications as directed. The contract will be non-enforceable, but it will provide patients with the opportunity to formally commit to a goal of taking the medications as prescribed. At 3 months, and 12 months, the participant will have the opportunity to reflect and modify adherence goals as desired.
  Other Names: Solid Organ Transplantation: An Educational Mini-Series for Patients
  Arms: Video education + adherence contract

SUMMARY:
This study aims to test the effectiveness of an electronic-based video intervention and behavioral contract on improving medication adherence among kidney transplant recipients.

DETAILED DESCRIPTION:
Non-adherence to immunosuppressive medications is a major problem after kidney transplantation, leading to increased rejections, hospitalizations and health care expenditures. Effective educational opportunities may positively influence adherence, especially when combined with a behavior intervention. However, increasing education and support to transplant recipients demands greater use of care providers' time and resources in a health care system that is already stretched.

A patient-oriented video series has been developed according to best practices for transplant education, featuring an animated character embarking on a transplant journey. Animated segments illustrate difficult concepts for patients with poor health literacy, and patient narratives provide support and encouragement. A multicenter randomized controlled trial will be conducted with 4 sites across North America. Patients will be randomized (1:1) to either the intervention (i.e., home-based video education + adherence contract plus usual care) or usual care alone. Patients will be enrolled in the study prior to hospital discharge and will be provided with access to the video intervention and contract electronically. The primary outcome will be adherence at 12 months post-transplant, as measured by self-report (BAASIS), and variability in immunosuppressant levels. Secondary outcomes include the change in knowledge score between the intervention and control in groups (measured by the Kidney Transplant Understanding Tool); differences in self-efficacy (Generalized Self-efficacy Scale), beliefs about medicines (Beliefs of Medicine Questionnaire), and quality of life (SF-12). Individualized viewing statistics will be analyzed to determine patient uptake, and satisfaction about the educational experience will be captured on a self-reported survey.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* can speak and understand and read English
* receive their first kidney transplant at one of the participating sites during enrolment

Exclusion Criteria:

* do not meet inclusion criteria
* have previously participated in a study entitle "Improving health outcomes of kidney recipients: A randomized controlled trial of a pre-transplant education intervention"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in adherence to immunosuppressant medications between intervention and control (self-report) | 3 months and 12 months after enrolment
  The Basel Assessment of Adherence to Immunosuppressive medications (BAASIS) will be sent electronically by self-reported survey. An answer of 'yes' to any of the questions (pertaining to missing doses, drug holidays, timing, and dose reduction) will constitute non-adherence as a binary outcome. • A continuous measure of adherence will also be determined in each individual using a visual analogue scale.
Difference in adherence to immunosuppressant medications between intervention and control (immunosuppressant blood levels) | 3 months and 12 months after enrolment
  Immunosuppressant levels (tacrolimus, cyclosporine or sirolimus) will be collected as per routine practice, and will be standardized to the patient specific target. Intra-patient coefficients of variation (CV) will be used as a measure of trough level variability, and percentage of sub-therapeutic levels will be determined for each patient.

SECONDARY OUTCOMES:
Difference in changes in kidney transplant knowledge between intervention and control | 3 months and 12 months after enrolment
  Measured by the Kidney Transplant Understanding Tool (K-TUT) via self-reported electronic survey. The K-TUT consists of 9 true/false and 13 multiple-choice questions, and scores are based on the number correct answers [YES/ NO format] of 69 items.
Difference in quality of life between intervention and control | 3 months and 12 months after enrolment
  Measured by the Short Form 12 (SF-12) via self-reported electronic survey. The SF-12 is a 12-item psychometric scale that measures functional health and well-being. Responses are indicated on a likert scale and aggregated into two sub scales; the mental component summary (MCS) and the physical component summary (PCS). The scores are converted to adjusted norm-based values of a healthy individual with a midpoint score of 50 indicating average health comparable to norm values.
Difference in self efficacy between intervention and control | 3 months and 12 months after enrolment
  Measured by the Generalized Self-Efficacy Scale (GSE) via self-reported electronic survey. The GSE measures an individual's self-beliefs in their ability to cope with various demands in life. It is a 10-item psychometric scale with a score for each item ranging from 1 to 4. The scores are summed and a higher score indicates stronger patient beliefs in self-efficacy.
Difference in education satisfaction between intervention and control | 3 months and 12 months after enrolment
  Measured by self-report electronic survey
Difference in beliefs about medication between intervention and control | 3 months and 12 months after enrolment
  Measured by the Beliefs of Medicine Questionnaire (BMQ) via self-reported electronic survey. The BMQ is an 18-item psychometric questionnaire which consists of two subscales. The BMQ-Specific assesses perceptions of medication prescribed for personal use, while the BMQ-General assesses beliefs about medications in general. The BMQ-General can be further classified into domain of General-Harm and General-Overuse. Items are scored on a 5-point likert scale, with higher score indicating stronger beliefs in each subscale.
Difference in adherence to transplant appointments between intervention and control | study end (12 months after enrolment)
  Captured by chart review
Video viewing habits (duration of viewing time) | study end (12 months after enrolment)
  We will record the total duration that participants have watched each video (in minutes). This number will be divided by the total length of each video and used as a surrogate marker for whether each video was watched in its entirety.
Cost of administering the intervention | study end (12 months after enrolment)
  Staff time and other resources used in administering the intervention will be tracked and monetized using market wages and prices.
Days in hospital | study end (12 months after enrolment)
  The number of days in hospital will be collected by chart review at the end of the study period to estimate health care utilization.

CONTACTS AND LOCATIONS:
Locations (3):
- University of Illinois Health Sciences System, Chicago, Illinois, United States
- Canada (2):
  - Southern Alberta Transplant Program, Calgary, Alberta
  - Saskatchewan Transplant Program, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Mansell H, Rosaasen N, Wichart J, West-Thielke P, Blackburn D, Liu J, Mainra R, Shoker A, Groot B, Wen K, Wong A, Bateni B, Luo C, Trivedi P. Video Education and Behavior Contract to Improve Outcomes After Renal Transplantation (VECTOR): A Randomized Controlled Trial. Patient Prefer Adherence. 2024 Jul 31;18:1589-1602. doi: 10.2147/PPA.S467142. eCollection 2024. PMID 39100428
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Mansell H, Rosaasen N, West-Thielke P, Wichart J, Daley C, Mainra R, Shoker A, Liu J, Blackburn D. Randomised controlled trial of a video intervention and behaviour contract to improve medication adherence after renal transplantation: the VECTOR study protocol. BMJ Open. 2019 Mar 13;9(3):e025495. doi: 10.1136/bmjopen-2018-025495. PMID 30872550
- See also: project website — https://words.usask.ca/transplant/
- See also: Vector protocol, BMJ open — https://bmjopen.bmj.com/content/9/3/e025495
- See also: Study Results — https://www.dovepress.com/video-education-and-behavior-contract-to-improve-outcomes-after-renal--peer-reviewed-fulltext-article-PPA